CLINICAL TRIAL: NCT02157207
Title: Racial and Aging Effects of Acute Antioxidant Supplementation
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Bo Fernhall, Dean, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2013-0980
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: antioxidants; Caucasians; healthy; African Americans; vascular; aging; racial differences
MeSH Terms: interventions — Antioxidants; Vitamin E; Ascorbic Acid; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be ingested in front of laboratory personnel in two doses, separated by 30 minutes to increase absorption, consumed 90 and 60 minutes before the testing protocol. Placebo microcrystalline cellulose capsules will be of similar taste, color and appearance.
  Interventions: Dietary Supplement: Antioxidant; Other: Placebo
- Antioxidant (Experimental): Supplementation will be ingested in front of laboratory personnel in two doses, separated by 30 minutes to increase absorption, consumed 90 and 60 minutes before the testing protocol. The first dose will consist of 300 mg of α-lipoic acid, 500 mg of vitamin C, and 200 IU of vitamin E, and the second dose will be 300 mg of α-lipoic acid, 500 mg of vitamin C, and 400 IU.
  of vitamin E.
  Interventions: Dietary Supplement: Antioxidant; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant — Comparison of antioxidant supplementation with a placebo. Effects of race and age and race in repsonse to the supplementation will be evaluated.
  Other Names: Vitamin E, Vitamin C, α-lipoic acid
Other: Placebo — Comparison of antioxidant supplementation with a placebo. Effects of race and age and race in repsonse to the supplementation will be evaluated.
  Other Names: No other names

SUMMARY:
This research is,being done to better understand how antioxidants (vitamins C, E and Alpha Lipoic Acid) af,f,ect the heart,and arteries. For this study, we will obtain blood samples to measure oxidative stress markers (substances in the blood that are linked to oxidative stress), cholesterol, insulin and blood glucose (sugar), as well as measure how well the heart and arteries are working following supplementation with the antioxidants.

Our central hypothesis is that acute antioxidant supplementation will improve arterial function at rest and during exercise in African Americans without an impact of age, whereas aging will modify these effects in Caucasians.

DETAILED DESCRIPTION:
The overall goal of this application is to investigate the effect of aging on how acute antioxidant supplementation affects decrements in arterial function observed in African Americans (AA). Additionally, this application will facilitate the applicant's emergence as an independent investigator in integrative clinical physiology. Oxidative stress (OS), contributes to hypertension, diabetes, heart failure, atherosclerosis, sepsis and aging. Increased OS leads to the development of endothelial dysfunction and subsequent development of cardiovascular disease through the inactivation of nitric oxide (NO) by superoxide (O2) and other free radicals. African Americans (AA) have increased OS and inflammation in vivo and in vitro, and have a lower serum concentration of most antioxidants. Endothelial cells of AAs have steady state NO/ O2/ONOO- balance that is close to redox state, which is a characteristic of endothelium impaired function disorders. Endothelium-derived NO is a vasodilator and inhibits monocyte adhesion and platelet activity and therefore is important in the maintenance of vascular homeostasis. These specific differences in OS could be a contributing mechanism to the high prevalence of cardiovascular disease, especially hypertension and heart failure, observed in AA. Aging causes increases in OS, endothelial dysfunction, and decreased arterial compliance, thus increasing the risk of cardiovascular disease. Acute supra-physiological dosages of antioxidants have been shown to transiently restore endothelial function in older adults and patients with coronary artery disease and hypertension by scavenging free radicals.However, it is unknown if acute antioxidant supplementation can diminish differences in vascular function between AA and Caucasians (CA). It is also unknown if acute antioxidant supplementation with known efficacy will differentially affect blood flow in AA vs CA during exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 or 55-75 years of age
* General Good health
* Without diagnosed atherosclerotic disease
* Without metabolic or inflammatory disease
* Do not use antioxidant vitamin supplementation
* Do not use anti-inflammatory medication within last 2 weeks
* Do not use steroidal substances within past 2 weeks
* Participants on medications (not listed in the Exclusion Criteria) will take medication as normal on all days of study visits.

Exclusion Criteria:

* Current smoker
* Severe obesity (BMI>40 kg/m2)
* Blood pressure greater than 140/90 mmHg
* Diabetes (fasting glucose >110 mg/dl)
* Hyperlipidemia (total cholesterol >240 mg/dl)
* Inflammatory disease (rheumatoid arthritis, systemic lupus erythematosus, etc)
* Diagnosed atherosclerotic heart disease
* Diagnosed cardiac arrhythmia
* Bacterial, viral or upper respiratory infection within past 1 month
* Bleeding disorder
* Anticoagulant medication
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 2 weeks
  The overall aim of this study is to examine the effects of an acute dose of an antioxidant cocktail on arterial stiffness (measured by ventral pulse wave velocity) in younger and older African Americans in comparison to younger and older Caucasians.
Arm blood flow | 2 weeks
  A second primary outcome is arm blood flow at rest and during two different intensities of hand grip exercise
Endothelial function | 2 weeks
  A third primary outcome is endothelial function assessed through brachial artery flow mediated dilation.

SECONDARY OUTCOMES:
Blood pressure | 2 weeks
  Both brachial and central blood pressure will be measured as secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fernhall, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois - Chicago, Chicago, Illinois, United States